CLINICAL TRIAL: NCT05982704
Title: Study of the Efficacy of Viral Neutralizing Monoclonal Antibodies Tiksagevimab/Cilgavimab and Regdanvimab for Omicron Strain Dominance in Patients With COVID-19
Brief Title: Study of Tixagevimab/Cilgavimab and Regdanvimab Efficacy for Treatment of COVID-19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: City Clinical Hospital No.52 of Moscow Healthcare Department (Other)
Collaborators: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Principal Investigator, Daria Fomina, Allergologist-immunologist, Head of the c Center of Allergy and Immunology, City Clinical Hospital No.52 of Moscow Healthcare Department
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05вн/0922
Record Dates: First submitted 2023-08-07; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Coronavirus Infections
Keywords: viral neutralizing monoclonal antibodies; Tixagevimab/Cilgavimab; Regdanvimab; Omicron strain
MeSH Terms: conditions — Coronavirus Infections | interventions — tixagevimab; regdanvimab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tixagevimab/cilgavimab (Group 1) (Experimental): tixagevimab/cilgavimab at a dose of 150+150 mg
  Interventions: Drug: tixagevimab/cilgavimab 150+150 mg
- tixagevimab/cilgavimab (Group 2) (Experimental): tixagevimab/cilgavimab at a dose of 300+300 mg
  Interventions: Drug: tixagevimab/cilgavimab 300+300 mg
- regdanvimab group (Active Comparator): regdanvimab at a dose of 40 mg/kg body weight
  Interventions: Drug: regdanvimab

INTERVENTIONS:
Drug: tixagevimab/cilgavimab 150+150 mg — Administration of tixagevimab/cilgavimab at a dose of 150+150 mg in patients with moderate/severe coronavirus infection.
  Other Names: EVUSHELD 150+150 mg
  Arms: tixagevimab/cilgavimab (Group 1)
Drug: tixagevimab/cilgavimab 300+300 mg — Administration of tixagevimab/cilgavimab at a dose of 300+300 mg in patients with moderate/severe coronavirus infection.
  Other Names: EVUSHELD 300+300 mg
  Arms: tixagevimab/cilgavimab (Group 2)
Drug: regdanvimab — Administration of regdanvimab at a dose of 40 mg/kg body weight in patients with moderate/severe coronavirus infection.
  Other Names: REGKIRONA
  Arms: regdanvimab group

SUMMARY:
Study hypothesis: the viral neutralizing monoclonal antibodies Tiksagevimab/Cilgavimab and Regdanvimab have high neutralizing activity against SARS-CoV-2 coronavirus, including Omicron strain, and may be effective in treating patients with moderate to severe COVID-19.

Description of the clinical study: Administration of monoclonal antibodies as antiviral therapy to patients with covid-19 and further Assesment of viral neutralizing monoclonal antibodies (Tiksagevimab/Cilgavimab and Regdanvimab) efficacy for treatment of new coronavirus infection (COVID-19) in adult patients. Participation of patients of both sexes aged 18 years or older with COVID-19 of moderate to severe course, hospitalized. Inclusion of 82 patients in the study: 38 in the tixagevimab/cilgavimab group (at a dose of 150+150 mg), 24 patients in the regdanvimab group (at a dose of 40 mg/kg body weight) and 20 patients in the tixagevimab/cilgavimab group (at a dose of 300+300 mg).

DETAILED DESCRIPTION:
Description of the intervention:

Hospitalized patients with moderate to severe coronavirus infection received three types of therapy: the tixagevimab/cilgavimab group (at a dose of 150+150 mg), the regdanvimab group (at a dose of 40 mg/kg body weight), and the tixagevimab/cilgavimab group (at a dose of 300+300 mg).

Further monitoring of the patient:

Screening period The screening period in the study begins with the signing of informed consent and lasts no longer than 24 hours (Visit 1, day 0) until the patient is included in the study (randomization).

Screening procedures:

* Obtaining informed consent.
* Collection of medical history (including previous COVID-19 history + dates; COVID-19 vaccination information + dates and type of vaccine used; revaccination data; data about co-morbidities as risk factors, etc.).
* Anthropometric data (height and weight) and demographic data.
* Physical exam.
* Collection of data on concomitant therapy.
* Assessment of vital signs: measuring blood pressure, pulse and body temperature, pulse oximetry (SpO2) and respiratory rate.
* Evaluation of SARS-CoV-2 virus test (smear PCR).
* CT scan of the lungs.
* Clinical blood count.
* Biochemical blood count.
* Complete urinalysis.
* ECG.
* Pregnancy test.
* Verification of eligibility for inclusion/inclusion.
* Decision of inclusion or exclusion of the patient.

Core period visits (drug prescription):

Visit 1 (Day 0-1) The conduct of Visit 1 takes place only after the patient has signed an informed consent form and the doctor-researcher has checked whether the inclusion/inclusion criteria are met)

* Blood sampling to determine the level of antigen-specific antibodies to SARS-CoV-2 and viral neutralizing activity of patients' blood sera against different variants of SARS-CoV-2 virus before drug using
* Sampling (nasal and oropharyngeal mucosa swabs) for PCR research or sequencing and viral load analysis
* Injection of the testing drug
* Interviewing the patient about subjective symptoms.
* Assessment of vital signs (BP, pulse and body tº measurements, pulse oximetry (SpO2) and frequency of breathing.
* ADR registration.
* Blood sampling to determine the level of antigen-specific antibodies to SARS-CoV-2 and viral neutralizing activity of patients' sera against different variants of SARS-CoV-2 virus immediately after administration testing drugs (Tixaghevimab/cilgavimab or Regdanvimab).

Visit 2 (Day 4)

* Physical exam.
* Collection of data on concomitant therapy.
* Assessment of vital signs: blood pressure, pulse and body tº measurements, pulse oximetry (SpO2) and frequency of breathing.
* Clinical blood count.
* Biochemical blood count.
* Sampling (nasal and oropharyngeal swabs) for PCR screening or sequencing and viral load analysis
* Blood sampling to determine the level of antigen-specific antibodies to SARS-CoV-2 and viral neutralizing activity of patients' sera against different variants of SARS-CoV-2 virus immediately after administration of the testing drugs (Tixaghevimab/cilgavimab or Regdanvimab).
* ADR registration.

Procedures for an unscheduled safety visit In case of clinical or laboratory signs of adverse reactions associated with the testing drug, an unscheduled visit should be scheduled. In addition to the scheduled emergency procedures and/or examinations, information on the combination therapy and adverse events is collected at the visit.

Minimum list of procedures for an unscheduled visit:

* Interviewing the patient about subjective symptomatology.
* Assessment of vital signs (BP, pulse and body tº measurements), pulse oximetry (SpO2) and frequency of breathing.
* Clinical blood count (may be ordered by the examining physician)
* Biochemical blood count (may be ordered by the examining physician)
* Registration and evaluation of ADR. Reporting to pharmacovigilance authorities (Roszdravnadzor) and to the pharmacovigilance department of the marketing authorization holder.

After the patient monitoring procedure, the efficacy and safety endpoints of the study drugs will be evaluated.

The volume of patients included in the study was formed on the basis of available resources and laboratory test capabilities related to efficacy endpoints of the investigational drugs, as well as clinical experience on the prescription of investigational drugs in scientific publications on this topic. After estimating the distribution of the sample, in the case of a non-normal distribution will be used nonparametric statistical methods for data analysis in IBM SPSS Statistics V.22. Numeric variables Numerical variables will be presented as medians and interquartile ranges (IQRs). Quantitative variables will be compared using Mann-Whitney U test and/or one-way Kruskal-Wallis analysis of variance. Fisher's exact test or χ2-square test will be used for qualitative variables. For all tests, p-value < 0,05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patient's signature of an informed consent form.
* Men and women aged 18 years or older.
* Confirmed diagnosis of new coronavirus infection COVID-19.
* Appearance of COVID-19 symptoms within 7 days prior to study inclusion
* Risk factors for COVID-19 progression and severity.

Exclusion Criteria:

* Patients with hypersensitivity to the active substance or other excipients (for the "Evusheld" product group: histidine, histidine hydrochloride monohydrate, sucrose, polysorbate 80, methionine; for the "Regkiron" product group: L-histidine, L-histidine monohydrate, polysorbate 80, L-arginine monohydrate)
* Patients with a history of anaphylactic reactions to drugs of monoclonal antibody class.
* Need for oxygen therapy at the time of study inclusion.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Viral neutralizing activity of patients' blood serum against different variants of SARS-CoV-2 virus (Wuhan and Omicron/ sublines BA.1, BA.2, BA.5) | On the first (0) day before the drug is administered; on the first day after the drug is administered; on the fourth day (4) after the drug is administered
  Preparation of serum samples for viral neutralizing activity analysis and determination of the level of viral neutralizing antibodies.
  Blood serum samples were inactivated at 56°C for 30 minutes in a solid-state thermostat. The neutralization reaction was performed in the constant dose-virus-serum dilution variant. Serum dilutions in DMEM culture medium with 2% inactivated fetal bovine serum were prepared, then 50 µl of serum dilutions were mixed with 100 TCID50 of SARS-CoV-2 virus (50 µl), incubated for 1 hour at 37°C and added to Vero E6 cells. The cells were incubated at 37ºC in 5% CO2, after 96 hours the cytopathic effect of the virus on the cell culture was recorded visually by assessing the disruption of the cell monolayer. The highest dilution of the tested serum, at which the cytopathic effect was suppressed, was taken as the viral neutralizing activity titer of the serum under study.
Viral load in nasopharyngeal swabs of patients by real-time PCR | On the first (0) day ; on the fourth day (4)
  Virus production, determination of infectious titer, and confirmation by PCR. Virus accumulation was performed in Vero E6 cells in DMEM medium with 2% inactivated FBS. The culture fluid containing the virus was aliquoted, frozen, and stored at -80C. The infectious virus titer was determined on Vero E6 cells by TCID50 determination. TCID50 titer was calculated using the Reed-Muench method.

SECONDARY OUTCOMES:
Adverse drug reaction | On the first day after the drug is administered; on the fourth day after the drug is administered; an unscheduled visit in event of an ADR
  Any medically adverse event detected in a patient or clinical trial subject after the use of a drug, which may or may not have a causal relationship to its use.
  The following information is given at the time of registration:
  * exact time of occurrence and resolution of the disorder
  * nature of the adverse event
  * severity (mild, moderate, severe)
  * Causal relationship to the study drug
  * Whether the adverse event is serious
  * Action taken (if ADR required treatment)
  * outcome
  * degree of expression

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow City Clinical Hospital 52, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Patient data will not be shared with other researchers due to the conditions of the study

REFERENCES:
- [Derived] Fomina DS, Lebedkina MS, Iliukhina AA, Kovyrshina AV, Shelkov AY, Andreev SS, Chernov AA, Dolzhikova IV, Kruglova TS, Andrenova GV, Tukhvatulin AI, Shcheblyakov DV, Karaulov AV, Lysenko MA, Logunov DY, Gintsburg AL. Real-world clinical effectiveness of Tixagevimab/Cilgavimab and Regdanvimab monoclonal antibodies for COVID-19 treatment in Omicron variant-dominant period. Front Immunol. 2023 Oct 20;14:1259725. doi: 10.3389/fimmu.2023.1259725. eCollection 2023. PMID 37928549